CLINICAL TRIAL: NCT02363933
Title: Phase II Feasibility Study to Evaluate the Efficacy and Safety of Perampanel in Seizure Patients With Primary Glial Brain Tumors
Brief Title: Perampanel in Seizure Patients With Primary Glial Brain Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00055609
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Brain Tumor, Primary
Keywords: Perampanel; Seizures
MeSH Terms: conditions — Brain Neoplasms; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perampanel + Current Anti-Epileptic Drug (Experimental): Primary glioma patients will receive perampanel along with their current AED for a total of 20 weeks. Perampanel will be titrated from 2 mg in weeks 1 and 2 and up to 8 mg daily by week 5 if well tolerated by the patient. They will then receive a maintenance dose of 8 mg per day through 16 weeks. After 16 weeks, subjects will be tapered off perampanel over a 4 week period.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel is a highly selective non-competitive alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) type glutamate receptor antagonist that has shown efficacy in a randomized phase III study for refractory partial-onset seizures
  Other Names: FYCOMPA

SUMMARY:
This is a Phase 2 single-arm study to assess the efficacy of perampanel as an adjunctive anti-epileptic drug (AED) in patients with primary glioma that are presenting refractory partial onset seizure activity (defined as 3 or more seizures in a 28-day period). In this study, patients will be started on a dose of 2 mg of perampanel daily taken orally at bedtime for 2 weeks. At the start of week 3 perampanel will be titrated up in dose in 2mg increments per week up to 8mg daily, as long as it is well tolerated by the patient. The highest dose of perampanel will be 8 mg orally at bedtime. Once this is achieved, patients will remain on a maintenance dose of 8 mg for 12 more weeks. The planned treatment dose is 8mg, but the dose can be modified by the physician based on patient reported tolerability. Titration and taper periods will be determined by the physician in the case where patients do not reach the planned treatment dose of 8 mg daily. Patients will be assessed in the Brain Tumor Center Clinic every 8 weeks. Study assessments will be made at enrollment, 8 weeks, 16 weeks, and 24 weeks. Assessments will include history and physical examination (H&P) including Karnofsky Performance Status (KPS), neurological examination, evaluation of seizure history, patient-reported outcomes of QoL, and computer based neurocognitive testing. After a total of 16 weeks of therapy, perampanel will be tapered down. At Week 17, patients will begin taking 6mg of perampanel, Week 18 4mg, Week 19 2mg, and Week 20 they will no longer take perampanel. Patients will be considered off treatment at the end of week 20, once perampanel has cleared their system. Patients will then be monitored through Week 24. Patients will continue to take their original AED regimen after they stop perampanel. If seizure control is achieved during the maintenance period or if seizures occur during the tapering period, patients can be continued on perampanel per the discretion of the treating physician. In this instance, perampanel will be prescribed by the treating physician and not provided within the confines of the study. Efficacy will be assessed using a log of patient-reported seizure activity. As is standard procedure at the Preston Robert Tisch Brain Tumor Center (PRTBTC), patients will be given a log to record the number of seizures that occur. Research team members will regularly contact patients for reminders and reports from the log. Safety will be assessed with the following laboratory evaluations: complete blood count (CBC) with differential, complete metabolic panel (CMP), and toxicity assessment.

DETAILED DESCRIPTION:
This is a Phase 2 single-arm study to assess the efficacy of perampanel as an adjunctive anti-epileptic drug (AED) in patients with primary glioma that are presenting refractory partial onset seizure activity (defined as 3 or more seizures in a 28-day period). In this study, patients will be started on a dose of 2 mg of perampanel daily taken orally at bedtime for 2 weeks. At the start of week 3 perampanel will be titrated up in dose in 2mg increments per week up to 8mg daily, as long as it is well tolerated by the patient. The highest dose of perampanel will be 8 mg orally at bedtime. Once this is achieved, patients will remain on a maintenance dose of 8 mg for 12 more weeks. The planned treatment dose is 8mg, but the dose can be modified by the physician based on patient reported tolerability. Titration and taper periods will be determined by the physician in the case where patients do not reach the planned treatment dose of 8 mg daily. Patients will be assessed in the Brain Tumor Center Clinic every 8 weeks. Study assessments will be made at enrollment, 8 weeks, 16 weeks, and 24 weeks. Assessments will include history and physical examination (H&P) including Karnofsky Performance Status (KPS), neurological examination, evaluation of seizure history, patient-reported outcomes of QoL, and computer based neurocognitive testing. After a total of 16 weeks of therapy, perampanel will be tapered for 3 weeks and then will be discontinued, such that Week 20 patients will no longer be taking perampanel. Patients will then be monitored through Week 24. Patients will continue to take their original AED regimen after they stop perampanel. Patients will remain on their original AED regimen during this treatment time and the dose of their original AED regimen at the start of the study will not be changed while they are on study. If seizure control is achieved during the maintenance period or if seizures occur during the tapering period, patients can be continued on perampanel per the discretion of the treating physician. In this instance, perampanel will be prescribed by the treating physician and not provided within the confines of the study. Efficacy will be assessed using a log of patient-reported seizure activity. As is standard procedure at the PRTBTC, patients will be given a log to record the number of seizures that occur. Research team members will regularly contact patients for reminders and reports from the log. Safety will be assessed with the following laboratory evaluations: complete blood count (CBC) with differential, complete metabolic panel (CMP), and toxicity assessment.

This study has been designed with 90% power to detect an increase in the 50% responder rate during the maintenance period from a benchmark of 20% to 35%. Assuming a type I error rate of 0.1, 61 patients will be required. Based on prior studies the early discontinuation rate was 16%, therefore 71 patients will be enrolled to compensate for patients discontinuing prior to the completion of the maintenance period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with a primary glioma and have refractory partial onset seizure activity (defined as 3 or more seizures in a 28-day period) on levetiracetam monotherapy
2. Adult patients (≥ 18 years old)
3. Karnofsky ≥ 70%
4. Hematocrit ≥ 29%, ANC ≥ 1,500 cells/L, platelets ≥ 100,000 cells/L
5. Serum creatinine ≤ 1.5 mg/dL, serum AST and bilirubin ≤ 1.5 times the upper limit of normal
6. If sexually active, patients will take contraceptive measures for the duration of protocol treatment and continue until two months after treatment. The effectiveness of hormonal contraceptives containing levonorgestrel has been shown to be reduced by perampanel at a 12 mg dose.1 Therefore, alternative or back-up methods of contraception are recommended.
7. Signed informed consent approved by the Duke Institutional Review Board

Exclusion Criteria:

1. Pregnant or breastfeeding (Both perampanel and other Anti-epileptic drugs are classified as Pregnancy Category C drugs.)
2. Chronic excessive use of psycho-pharmaceuticals, alcohol, illicit drugs, or narcotics
3. Inability to complete or perform measures of patient-reported outcomes or neurocognitive testing on the computer
4. Known allergy to perampanel
5. Concomitant use of known cytochrome P450 inducers such as carbamazepine, phenytoin, or oxcarbazepine (see Appendix A)
6. Previous history of suicidal ideation, homicidal ideation, depression leading to hospitalization or mood disturbance leading to hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject decided not to participate-had no more seizures after enrolling/while waiting to start
Period: Overall Study
Arm/Group | Perampanel + Current Anti-Epileptic Drug
Started | 8
Completed | 2
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Perampanel + Current Anti-Epileptic Drug
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With ≥50% Seizure Reduction During the Maintenance Period Compared With Seizure Frequency Before Initiation of Perampanel
Description: The primary objective of this study is to assess the efficacy of perampanel as an adjunctive anti-epileptic drug (AED) in patients with primary glioma presenting refractory partial onset seizure activity. Efficacy will be assessed by the 50% responder rate, defined as the percentage of patients with a ≥50% seizure reduction during the maintenance period compared with the seizure frequency before initiation of perampanel. Seizure frequency during maintenance perampanel will be computed as the ratio of the total number of seizure episodes while receiving perampanel during the maintenance period and the number of days perampanel is administered
Time Frame: 20 Weeks
Population: Seizure frequency was not systematically gathered at screening. As the 50% responder rate requires an adequate baseline comparison, it is not possible to compute the 50% responder rate.
Arm/Group | Perampanel + Current Anti-Epileptic Drug
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Patients Who Experience a Adverse Event Possibly, Probably, or Definitely Attributable to Perampanel Treatment
Description: The percentage of patients with unacceptable adverse events that are possibly, probably, or definitely related to perampanel treatment will be calculated. Unacceptable adverse events include all Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 Grade 4 or 5 toxicities that are possibly, probably, or definitely related to perampanel, as well as suicidal ideation (any grade) or suicide attempt (Grade 3-5).
Time Frame: 24 Weeks
Population: All patients treated with perampanel is included in the attributable adverse event rate.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel + Current Anti-Epileptic Drug
Number analyzed (Participants) | 8
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Perampanel + Current Anti-Epileptic Drug
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel + Current Anti-Epileptic Drug (N=8)
Multi-organ failure (General disorders) | 1
Lung infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel + Current Anti-Epileptic Drug (N=8)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Mucosal infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Anemia (Investigations) | 1
Anmia (Investigations) | 1
Creatinine increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Pyramidal tract syndrome (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02363933/Prot_SAP_000.pdf